CLINICAL TRIAL: NCT00925483
Title: Decreasing Dialysis Cardiovascular Risk: Daily Versus Longer Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Devasmita Dev MD, Dallas VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #04-050
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Cardiovascular Disease
Keywords: left ventricular mass; cardiac MRI; long dialysis; daily dialysis
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- daily long (Experimental): daily long (4 hours, 6 times weekly) dialysis for 6 months
  Interventions: Procedure: dialysis
- daily short (Experimental): daily short (2 hours 6 times weekly) dialysis for 6 months
  Interventions: Procedure: dialysis
- alternate day conventional (Experimental): alternate day conventional (4 hours, 3 times weekly) dialysis for 6 months
  Interventions: Procedure: dialysis
- alternate day long (Experimental): alternate day long (8 hours, 3 times weekly) dialysis for 6 months
  Interventions: Procedure: dialysis

INTERVENTIONS:
Procedure: dialysis — different dialysis schedules for each arm

SUMMARY:
Given the known increased risk of heart disease in hemodialysis patients, this study aims to evaluate the change in both size and function of the heart by using cardiac magnetic resonance imaging (MRI) in patients undergoing either daily long (4 hours, 6 times weekly), daily short (2 hours 6 times weekly), or alternate day conventional (4 hours, 3 times weekly) and alternate day long (8 hours, 3 times weekly) dialysis for 6 months from randomization. The patients are randomly put in the groups based on predetermined randomization schedule and the cardiologist trained in cardiac MRI readings is blinded to the patient treatment schedule. Given that changes in heart function may be seen with cardiac imaging techniques within 6 months, the expectation is that groups on daily treatment may have better outcome for this parameter as changes in volume and blood pressure may also be affected in a positive way in patients on daily dialysis.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease patients on hemodialysis

Exclusion Criteria:

* Weight > 350 lbs
* Known poor dialysis and or treatment compliance
* Unable to come for daily treatments if randomization occurs in this group
* Prognosis less than 6 months
* Difficulty in tolerating dialysis and possibility of discontinuation of dialysis before 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-08; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
LVM change per Cardiac MRI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Devasmita C. Dev, MD, Principal Investigator — VA North Texas Health Care System, Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States